CLINICAL TRIAL: NCT01023945
Title: A Phase 1, Randomized, Double-blind, Placebo Controlled, Monotherapy Study to Assess the Pharmacodynamics, Pharmacokinetics, Safety and Tolerability of ASP1941 in Japanese Patients With Type 2 Diabetes Mellitus
Brief Title: A Study of ASP1941 in Japanese Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1941-CL-0070
Record Dates: First submitted 2009-11-30; First posted 2009-12-02 (Estimated); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: ASP1941; Diabetes mellitus; Blood glucose
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — ipragliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- ASP1941 high dose group (Experimental): oral
  Interventions: Drug: ASP1941
- ASP1941 low dose group (Experimental): oral
  Interventions: Drug: ASP1941
- Placebo group (Placebo Comparator): oral
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASP1941 — oral
  Arms: ASP1941 high dose group; ASP1941 low dose group
Drug: Placebo — oral
  Arms: Placebo group

SUMMARY:
The primary purpose of this study is to evaluate the pharmacodynamic profile (blood glucose and urinary glucose excursion) of ASP1941 in patients with type 2 diabetes mellitus. Safety, tolerability and pharmacokinetics are also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients for at least 12 weeks
* HbA1c value between 7.0 and 10.0% at screening
* Fasting plasma glucose ≥ 126mg/dL and < 240mg/dL at screening
* Body Mass Index (BMI) 20.0 - 45.0 kg/m2.

Exclusion Criteria:

* Type 1 diabetes mellitus patients
* Serum creatinine > upper limit of normal
* Proteinuria（albumin/creatinine ratio > 300mg/g）
* Dysuria and/or urinary tract infection
* Significant renal, hepatic or cardiovascular diseases
* Severe gastrointestinal diseases

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-11-07 (Actual); Primary Completion 2010-03-26 (Actual); Study Completion 2010-03-26 (Actual)

PRIMARY OUTCOMES:
Change in plasma glucose levels | On day 14

SECONDARY OUTCOMES:
Urinary glucose excursion | On day 14
Pharmacokinetic parameter of ASP1941 | On day 14
Safety by adverse events, routine safety laboratories and vital signs. | During treatment
Change in serum insulin levels | On day 14

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (1):
- Kantou, Japan

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Toyoshima J, Saito M, Kaibara A, Isaka H, Sakatani T. Comparison of the Pharmacokinetic and Pharmacodynamic Relationship of Ipragliflozin Between Patients With Type 1 and Type 2 Diabetes Mellitus. Clin Ther. 2020 Sep;42(9):1787-1798.e3. doi: 10.1016/j.clinthera.2020.07.009. Epub 2020 Aug 21. PMID 32839028
- See also: Link to results on Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=90